CLINICAL TRIAL: NCT04769427
Title: Non-Surgical Rhinoplasty Using Polydioxanone Threads
Brief Title: Non-Surgical Rhinoplasty Using PDO Threads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PDO-122020
Record Dates: First submitted 2021-01-20; First posted 2021-02-24 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Nasal Defect

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PDO Max thread injection to nose (Experimental)
  Interventions: Device: PDO max threads

INTERVENTIONS:
Device: PDO max threads — To determine the effects of absorbable Polydioxanone (PDO) thread non-surgical rhinoplasty on quality of life (FACE-Q scale)

SUMMARY:
To determine the effects of absorbable Polydioxanone (PDO) thread non-surgical revision rhinoplasty on first impressions and quality of life (FACE-Q scale) in 10 patients who desire further changes to their nasal tip and/or nasal dorsum

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of ages 18 and above.
2. Subjects will be required not to have had previous filler injections, or other cosmetic treatments to the nose within the last 12 months.
3. Subjects that understand the purpose and aspects of the study, freely sign the consent and complete the required treatment and follow up visit.

Exclusion Criteria:

1. Males and females below age of 18.
2. Subjects who have had previous surgery, filler injections, or other cosmetic treatments to the nose within the last 12 months.
3. Patients with any prior nasal implants
4. Subjects who are pregnant or nursing.
5. Subjects with a known allergy or sensitivity to any component of the study ingredients.
6. Any history of bleeding disorders (iatrogenic or otherwise). This includes persons who have undergone therapy with thrombolytics, anticoagulants, or inhibitors of platelet aggregation in the preceding 3 weeks.
7. Anyone taking aspirin, ibuprofen, St. John's Wort, or high doses of Vitamin E supplements in the last 3 weeks.
8. Subjects with diseases, injuries, or disabilities of the nose, including those with autoimmune disease affecting the nose
9. Subjects that do not understand the purpose and aspects of the study, do not sign the consent and do not complete the required treatment and follow up visit will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Non -surgical rhinoplasty using PDO Max threads | 1 month
  The effects of absorbable Polydioxanone (PDO) thread non-surgical rhinoplasty on quality of life (FACE-Q scale). FACE-Q scales are rated from 1-4 with ratings closer to 4 as more favorable.

SECONDARY OUTCOMES:
Non -surgical rhinoplasty using PDO Max threads | 1 month
  The effects of absorbable Polydioxanone (PDO) thread non-surgical rhinoplasty on first impressions (using the first impression questionnaire). Questionnaire is rated from 1 to 10 with results closer to 10 as more favorable.
Non -surgical rhinoplasty using PDO Max threads | 1 month
  The efficacy in reduction of nasal dorsum convexity, and improvement of tip rotation and projection as measured on pre/post injection 2D photographs

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States